CLINICAL TRIAL: NCT00668135
Title: Randomised, Double Blind, Placebo Controlled, Parallel Group, Multi-centre, Multinational Study to Evaluate the Efficacy and Tolerability of Vardenafil (BAY 38-9456) in Treatment of Male Erectile Dysfunction in Asia
Brief Title: Assessment of Vardenafil in Patients With Erectile Dysfunction in Asia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10657
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Vardenafil (Levitra, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil (Levitra, BAY38-9456) — Vardenafil 10 mg orally on demand prior to intercourse
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
To demonstrate the efficacy, safety and tolerability of 10 mg oral vardenafil (BAY 38-9456) compared to placebo for a period of 12 weeks in men with erectile dysfunction (ED)

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 years and older- Males with erectile dysfunction
* Stable heterosexual relationship Exclusion Criteria:
* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months- Nitrate use
* Other exclusion criteria apply according to the Summary of Product Characteristics

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2003-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF) Questionnaire and Sexual Encounter Profile question 2 (SEP 2) and Sexual Encounter Profile question 3 (SEP 3) | 12 weeks

SECONDARY OUTCOMES:
Global Assessment Question | 12 weeks
Other diary responses | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Hong Kong, Hong Kong
- Jakarta, Jakarta Special Capital Region, Indonesia
- Malaysia (3):
  - Petlaing Jaya, Salangor
  - Kuching, Sarawak
  - Kuala Lumpur
- Manila, Philippines
- Singapore, Singapore
- Bangkok, Bangkok, Thailand